CLINICAL TRIAL: NCT07148752
Title: Evaluation of Amoebicidal Efficacy of Resveratrol and Resveratrol Loaded Nanoparticles on Acanthamoeba Keratitis Isolates
Brief Title: Evaluation of Resveratrol and Its Loaded Nanoparticles on Acanthamoeba
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Hany Mohammed, assistant lecturere, Assiut University
Other Study IDs: Acanthamoeba new treatment
Record Dates: First submitted 2025-08-11; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Corneal Ulcer Caused by Acanthamoeba

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Acanthamoeba is a free-living amoeba responsible for severe human infections. There are at least twenty-two different genotypes of Acanthamoeba (T1-T22). T4 is the most common virulent genotype, mainly Acanthamoeba castellani and Acanthamoeba polyphaga.

Proper treatment still represents a challenge for healthcare professionals.So, we need novel therapeutic strategies, including newer drugs and/or drug delivery systems that can overcome the developing drug resistance as well as have minimal toxicity to human cells.

There is a new approach in the treatment of parasitic disease by using nanotechnology and natural compounds as plant extracts.

The current study aims to evaluate the therapeutic potential of resveratrol, both in its free form and when loaded on nanoparticles, against clinically isolated Acanthamoeba strains obtained from patients with persistent AK or corneal ulcers.

DETAILED DESCRIPTION:
: 1-Specimen collection using: A- Corneal swabs. B- Corneal scraping and superficial keratectomy.

C- Contact lenses and contact lens solutions. 2-Culture: The collected samples will be cultivated on non-nutrient agar (NNA) plates seeded with heat-killed Escherichia coli.

3-Cultivation and maintenance of Acanthamoeba isolates in axenic culture: PYG media will be used in order to obtain a significant number of parasites with a minimum presence of bacteria.

4-Molecular analysis:Positive samples by culture will be subjected to conventional PCR technique for molecular characterization of Acanthamoeba at the genus level using genus-specific primers: Forward primer JDP1: F5'-GGC CCAGATCGTTTACCGTGAA-3'

- Reverse primer JDP2:R5' TCTCACAAGCTGCTAGGG AGTCA-3' 5- Sequencing and phylogenetic study: The amplified DNA will be purified, sequencing ASA.S1 region of the 18s rRNA gene will be performed. Following genotyping, the Basic Local Alignment Search Tool (BLAST) of the US National Center for Biotechnology Information (NCBI) will be used to identify similar Acanthamoeba sequences.

6-Experimental study: Preparation of Resveratrol (Plant extract), preparation and Characterization of nanoparticles and parasite material preparation from PYG axenic culture media will be done.

study groups: Group 1: Negative control: No drug is applied. Group 2: Positive control: Propamidine isethionate as a reference drug. Group 3: Resveratrol alone is applied. Group 4: Nanoparticles alone are applied. Group 5: Resveratrol loaded nanoparticles.

* Group 6: Propamidine isethionate and Resveratrol.
* Group 7: Propamidine isethionate and Resveratrol loaded nanoparticles.

I- In-vitro experimental study:

For assessment of applied drugs/extracts efficacy:

A- In vitro drug susceptibility testing :The Acanthamoeba isolates will be tested for their susceptibility to various drug groups serial dilutions. The number of cysts/trophozoites will be counted using a hemocytometer.

B-Viability measurements: Using trypan blue viability stain. C-Scanning electron microscopy (SEM) D-Host cells cytotoxicity evaluation using MTT assay on HeLa cell line: The MTT assay (3-[4,5-dimethylthiazol-2-yl]-2,5-diphenyl tetrazolium bromide) will be performed to determine the cell cytotoxicity of the tested extract on human cells that are represented by the HeLa cell line.

-Percentage of cell cytotoxicity will be calculated, and the acceptable limit of cytotoxicity will be taken as the viability cutoff of 60%; thus, a cytotoxicity of >40% is considered unacceptable.

II- In-vivo experimental study:

-Sample size calculation: The sample size is calculated to be 35 tested animals (5 in each group).

* Procedure:

  1. Induction of keratitis and confirmation of the infection
  2. Application of the tested drug (7 groups as previously discussed).
* Evaluation of treatment by:

  1. Clinical evaluation (examination and scoring of the tested animal's eyes).
  2. Histopathological evaluation of the animal's corneal tissue:
  3. Parasitological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presented with keratitis to the outpatient clinic.
2. Patients presented with corneal ulcers to the outpatient clinic.

Exclusion Criteria:

1. Patients presented with corneal ulcers caused by pathogens rather than Acanthamoeba (bacterial, viral or fungal).
2. Patients presented with other eye conditions that act as confounding variable as corneal perforation, severe dry eye, glaucoma, scleritis and active uveitis.
3. Patients with history of previous ocular surgery or corneal transplant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: study participants will be enrolled form Ophthalmology department clinics
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Invitro evaluation of amoebicidal efficacy of resveratrol and resveratrol loaded nanoparticles against the isolated Acanthamoeba pathogenic strains from corneal ulcers patients in comparison to the reference drug through experimental study. | 2025-2028
  In-vitro experimental study:
  A-Drug susceptibility testing :The Acanthamoeba isolates will be tested for their susceptibility to various drug groups serial dilutions. The number of cysts/trophozoites will be counted using a hemocytometer.
  B-Viability measurements: Using trypan blue viability stain. C-Scanning electron microscopy (SEM).
  D-Host cells cytotoxicity evaluation using MTT assay on HeLa cell line:
  -Percentage of cell cytotoxicity will be calculated, and the acceptable limit of cytotoxicity will be taken as the viability cutoff of 60%; thus, a cytotoxicity of >40% is considered unacceptable.
Invivo evaluation of amoebicidal efficacy of resveratrol and resveratrol loaded nanoparticles against the isolated Acanthamoeba pathogenic strains from corneal ulcers patients in comparison to the reference drug through experimental study. | 2025-2028
  II- In-vivo experimental study:
  * The sample size is calculated to be 35 tested animals (5 in each group).
  * Procedure:
  Induction of keratitis and confirmation of the infection Application of the tested drug (7 groups as previously discussed).
  -Evaluation of treatment by: Clinical evaluation (examination and scoring of the tested animal's eyes).
  Histopathological evaluation of corneal tissue:
  Parasitological evaluation.

IPD SHARING:
Plan to Share IPD: No